CLINICAL TRIAL: NCT04315961
Title: Effects of Dietary Conditions on Drug Response
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit participants.
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00231935; R01DA003890 (NIH)
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: over-the-counter; prescription medication; subjective effects

STUDY DESIGN:
Intervention Model Description: This is a within-subjects design. This study involves administration of drug conditions in different dose sequence orders. All participants will receive the same drug conditions, but the order in which the participants receive the drug conditions will be different across participants. Participants will be randomly assigned to one of several different dose sequences. As part of instructions during the informed consent process, volunteers will be given a list of drugs volunteers may receive rather than informing volunteers only of the specific drugs being administered. More drugs are listed than will be administered to increase the degree to which volunteers are "blind" to the drugs being studied. Researchers will be blind to the drug conditions on any given session because a pharmacy member with no participant interaction will assign the randomized dose sequence and prepare the study drugs.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Please note: This is a double-blind study. As part of instructions during the informed consent process, volunteers will be given a list of drugs volunteers may receive rather than informing volunteers only of the specific drugs being administered. More drugs are listed than will be administered to increase the degree to which volunteers are "blind" to the drugs being studied. Researchers will be blind to the drug conditions on any given session because a pharmacy member with no participant interaction will assign the randomized dose sequence and prepare the study drugs. Masking:Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Caffeine Maintenance (Experimental): All participants will receive the same drug conditions, but the order in which the participants receive the drug conditions will be different across participants. Thus, comparisons of the drug conditions on mood and choice will be compared within-subjects (e.g., between drug and placebo). During the caffeine maintenance condition, participants will ingest 200 mg of caffeine orally in capsules three times daily.
  Interventions: Drug: Blinded drug dose conditions
- Placebo Maintenance (Placebo Comparator): All participants will receive the same drug conditions, but the order in which the participants receive the drug conditions will be different across participants. Thus, comparisons of the drug conditions on mood and choice will be compared within-subjects (e.g., between drug and placebo). The placebo maintenance condition will be identical to the caffeine maintenance condition, with the exception that the thrice daily capsules will contain placebo (microcrystalline cellulose) rather than containing caffeine.
  Interventions: Drug: Blinded drug dose conditions

INTERVENTIONS:
Drug: Blinded drug dose conditions — Capsules will contain commonly prescribed or over-the-counter drugs or placebo. Capsules in this study may contain sedatives, muscle relaxants, or anti-anxiety medications, stimulant drugs/weight loss medications, or antihistamines which must remain blinded for the purposes of this study.

SUMMARY:
This non-treatment study will examine how different dietary conditions may affect a person's response to commonly used drugs.

DETAILED DESCRIPTION:
Volunteers (aim is 36 completers) will participate in a double-blind study conducted over a period of about 10-12 weeks including sessions for screening, food and beverage diary review, and drug exposure sessions. During screening, participants will be asked questions about participants' general characteristics including demographic information, mood, and personality. Participants will also be examined to determine medical eligibility. Eligible participants will complete diary sessions (4 total), experimental sessions (12 total) and end of study sessions (2 sessions). At food diary sessions, participants will be asked to eliminate certain foods and beverages from participants' diet, record daily food and beverage consumption and attend the laboratory approximately two times to discuss participants' food diaries. At these sessions, participants will orally ingest capsules containing commonly prescribed medications, over-the-counter medications, and/or placebo and will receive study capsules in blister packs which participants will take three times daily throughout the study. During experimental sessions, food and beverage restrictions will remain in place, participants will continue thrice daily capsule administration and will also be exposed to experimental test sessions. Participants will report to the laboratory 2-3 times weekly in order to ingest study capsules, receive blister packs and fill out questionnaires. After leaving the laboratory, participants will be asked to fill out surveys remotely in order to describe the effects of that session's capsules on mood and preference. After completing the first six sessions, participants will receive a mid-study bonus and have a 1-week break from attending sessions, during which participants will continue to swallow capsules thrice daily. Participants will return to the lab and complete two food diary sessions. After this, participants will complete experimental test sessions 7-12, where participants will again swallow capsules and complete questionnaires. After completing experimental test sessions 1-12, participants will complete a final experimental test session to facilitate the study assessment of subjective monetary value of drug conditions. Finally, participants will return to the laboratory to receive a bonus payment for study completion and to complete an end-of-study questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Fluent in written and spoken English and is capable of understanding and complying with the protocol
* Medically healthy
* Non-smoker
* Appropriate dietary/over-the-counter/prescription/illicit drug use history
* Body Mass Index between 18.5 and 34.9
* Appropriate use of birth control in females e.g., barrier methods, hormonal contraceptives, Intra Uterine Devices (IUDs)

Exclusion Criteria:

* Known hypersensitivity to administered drugs
* Current neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary or metabolic disease for which administration of the study drugs would be contraindicated
* Current psychiatric or substance use condition that would interfere with study participation
* Diastolic blood pressure >90 mmHg or a systolic pressure of >140 mmHg
* Use of medications that would interfere with study participation
* Unwilling or unable to comply with the protocol
* Any other serious disease or condition that might affect life expectancy or make it difficult to successfully manage the subjects according to the protocol
* Females: Pregnancy, breastfeeding, or plans to become pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Sweeney, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is not currently a plan to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Within-Subjects Dose Conditions: All participants will receive the same drug conditions, but the order in which the participants receive the drug conditions will be different across participants. Thus, comparisons of the drug conditions on mood and choice will be compared within-subjects (e.g., between drug and placebo) and not between arms.
  Blinded drug dose conditions: Capsules will contain commonly prescribed or over-the-counter drugs or placebo. Capsules in this study may contain sedatives, muscle relaxants, or anti-anxiety medications, stimulant drugs/weight loss medications, or antihistamines which must remain blinded for the purposes of this study.
Period: Overall Study
Arm/Group | Within-Subjects Dose Conditions
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Within-Subjects Dose Conditions
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: Peak Participant Subjective Ratings of Drug Liking
Description: Primary outcome will be peak change in participant ratings of drug liking relative to pre-drug ratings within 4 hours post-administration during experimental test sessions. Participants rate drug liking on a scale from -4 (dislike very much) to 4 (like very much) where 0 = Neutral or No Effect. This is not a treatment study, and higher or lower ratings of drug liking do not represent better or worse outcomes.
  The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Up to 4 hours after capsule ingestion during experimental test session
Population: as for baseline characteristics
Arm/Group | Within-Subjects Dose Conditions
Number analyzed (Participants) | 0

2. Secondary Outcome: Participant Subjective Ratings of Drug Value
Description: Secondary outcome will be subject rating of monetary drug value as assessed post-administration during experimental test sessions. Participants will rate the subjective value of the drug on a scale from -$30 (i.e., they would prefer to lose $30 rather than take the drug) to $30 (i.e., they would prefer to take today's drug instead of receiving $30). This is not a treatment study, and higher or lower ratings of drug value do not represent better or worse outcomes.
  The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Up to 4 hours after capsule ingestion during experimental test session
Population: as for baseline characteristics
Arm/Group | Within-Subjects Dose Conditions
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Within-Subjects Dose Conditions
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination - Study was terminated due to COVID 19 lockdown and subsequent research restrictions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04315961/Prot_SAP_000.pdf